CLINICAL TRIAL: NCT04779645
Title: The Effects of Glucagon Antagonism on Insulin Sensitivity, Cardiovascular Risk, and Ketogenesis in Type 1 Diabetes
Brief Title: Effects of GRA in Patients With Type 1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: REMD Biotherapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Jeremy Pettus, MD, Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UC-MEDJP-04
Record Dates: First submitted 2021-02-22; First posted 2021-03-03 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — volagidemab

STUDY DESIGN:
Intervention Model Description: Single-center, double-blind, placebo-controlled, multi-dose study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GRA (REMD-477) Group (Experimental): Once weekly, subcutaneous injection of 70mg REMD-477 (in 1 mL solution) for up to 12 weeks.
  Interventions: Drug: REMD-477
- Placebo Group (Placebo Comparator): Once weekly, subcutaneous injection of 1mL saline solution for up to 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REMD-477 — 12-Week, once weekly subcutaneous injection with 70mg REMD-477
  Arms: GRA (REMD-477) Group
Drug: Placebo — 12-Week, once weekly subcutaneous injection with placebo
  Arms: Placebo Group

SUMMARY:
This study will examine the effects a Glucagon Receptor Antagonist (GRA), has on Insulin Sensitivity, Cardiovascular risks (CVD), and Ketone body formation in participants with Type 1 diabetes. The participants will complete blood tests, tests to measure energy expenditure, CVD risks, and insulin resistance. These tests will be performed prior to start of treatment and again after 12-weeks of treatment with the GRA (called REMD-477).

DETAILED DESCRIPTION:
This single-center, double-blind, placebo-controlled, multi-dose study is designed to evaluate the effects of glucagon antagonism on insulin sensitivity, cardiovascular risk and ketogenesis in individuals with Type 1 Diabetes. To accomplish the specific aims proposed, a single clinical trial will be conducted in which a maximum of 30 subjects with T1D, who are otherwise healthy, will be treated with REMD-477 or matching placebo for up to 12 weeks at a dose of 70mg (administered subcutaneously each week) with assessments done pre- and post-therapy. Subjects will be randomized on a 1:1 basis to either the REMD-477 group or placebo group and all subjects will remain on their standard of care insulin therapy throughout the study. There will be 19 study visits as outlined below:

1. Screening - Complete consenting process, complete medical history and physical exam, review of current medications, collect height/weight, vital signs, and fasting laboratory (blood and urine) tests.
2. Baseline Visit 1 - Participants that meet screening criteria will complete cardiovascular tests including flow mediated dilation and EndoPat, complete vital signs, weight and laboratory tests for safety and CVD markers.
3. Baseline Visit 2 - Participants will complete a 2-Step Hyperinsulinemic/Euglycemic clamp with tracer, Indirect Calorimetry, muscle and adipose tissue biopsies.
4. Baseline Visit 3 - Insulin withdrawal challenge and injection #1 of REMD-477 or placebo. Participants will suspend insulin delivery and remove insulin pump. Blood sugars and ketones will be monitored for up to 8 hours.
5. Visit 4 - Injection #2 of REMD-477 or placebo and blood collection for safety labs.
6. Visit 5 - Injection #3 of REMD-477 or placebo.
7. Visit 6 - Injection #4 of REMD-477 or placebo and blood collection for safety labs.
8. Visit 7 - Injection #5 of REMD-477 or placebo.
9. Visit 8 - Injection #6 of REMD-477 or placebo and blood collection for safety labs.
10. Visit 9 - Injection #7 of REMD-477 or placebo.
11. Visit 10 - Injection #8 of REMD-477 or placebo and blood collection for safety labs.
12. Visit 11 - Injection #9 of REMD-477 or placebo.
13. Visit 12 - Injection #10 of REMD-477 or placebo and blood collection for safety labs.
14. Visit 13 - Injection #11 of REMD-477 or placebo.
15. Visit 14 - Injection #12 of REMD-477 or placebo and blood collection for safety labs.
16. Visit 15 - Repeat cardiovascular tests including flow mediated dilation and EndoPat, complete vital signs, weight and laboratory tests for safety and CVD markers.
17. Visit 16 - Repeat 2-Step Hyperinsulinemic/Euglycemic clamp with tracer, Indirect Calorimetry, muscle and adipose tissue biopsies.
18. Visit 17 - Repeat Insulin withdrawal challenge. Participants will suspend insulin delivery and remove insulin pump. Blood sugars and ketones will be monitored for up to 8 hours.
19. Visit 18 - Safety follow-up visit that includes physical exam, vitals, blood and urine sample collection.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 18 and 65 years old, inclusive, at the time of screening;
2. Females of non-child bearing potential must be ≥ 1 year post-menopausal or documented as being surgically sterile. Females of child bearing potential must agree to use two methods of contraception during the entire study and for an additional 3 months after the end of dosing with the investigational product;
3. Male subjects must be willing to use clinically acceptable method of contraception during the entire study and for an additional 6 months after the end of the treatment period;
4. Diagnosed with Type 1 diabetes based on clinical history or as defined by the current American Diabetes Association (ADA) criteria for > 5 years;
5. Treatment with a stable insulin regimen for at least 8 weeks before screening with continuous subcutaneous insulin infusion (CSII) via an insulin pump;
6. Currently using a Continuous Glucose Monitoring (CGM) system;
7. HbA1c ≤ 8.5 % at screening;
8. A minimum weight of 50kg;
9. eGFR ≥ 60 mL/min/1.73m²
10. Able to provide written informed consent approved by an Institutional Review Board (IRB).

Exclusion Criteria:

1. History or evidence of clinically-significant disorder or condition that, in the opinion of the Investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion;
2. History of pancreatitis, medullary thyroid carcinoma and/or liver disease;
3. Clinically significant diagnosis of anemia;
4. Body Mass Index (BMI) < 18.5 kg/m2 and/or weight less than 50kg;
5. Whole blood donation of 1 pint (500 mL) within 8 weeks prior to Screening. Donations of plasma, packed RBCs, platelets or quantities less than 500 mL are allowed at investigator discretion;
6. Current or recent (within 1 month of screening) use of diabetes medications other than insulin;
7. Women who are pregnant or lactating/breastfeeding;
8. Unable or unwilling to follow the study protocol or who are non-compliant with screening appointments or study visits;
9. Any other condition(s) that might reduce the chance of obtaining study data, or that might cause safety concerns, or that might compromise the ability to give truly informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-31 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Metabolic Clearance Rate of Insulin | 12-Weeks
  The change from baseline in calculated metabolic clearance rate of insulin as measured by the 2-step Hyperinsulinemic-Euglycemic Clamp.
Rate of Resting Energy Expenditure (REE) | 12-Weeks
  Change from baseline REE as measured by indirect calorimetry.
Change in Beta-hydroxybutyrate (BHB) Level | 12-Weeks
  The change from baseline in peak BHB production as measured by the insulin withdrawal challenge.
Change in Free Fatty Acid (FFA) Level | 12-Weeks
  The change from baseline in peak FFA production as measured by the insulin withdrawal challenge.
Change in mRNA Expression | 12-Weeks
  The change from baseline in gene mRNA expression as measured by adipose and muscle tissue samples.
Change in Peripheral Macrovascular Vasodilation | 12-Weeks
  The change from baseline in post-stimulus vessel diameter as measured by flow mediated dilation.
Change in Peripheral Microvascular Vasodilation | 12-Weeks
  The change from baseline in reactive hyperemia index as measured by reactive hyperemia-peripheral arterial tonometry (RH-PAT).
Change in Cardiovascular Disease (CVD) Risk Markers. | 12-Weeks
  The change in pg/mL from baseline in CVD risk markers (SAA, CRP, VCAM-1 and ICAM-1) as measure by blood samples.
Change in Cardiovascular Disease (CVD) Risk Markers. | 12-Weeks
  The change in ng/mL from baseline in CVD risk markers (Thrombomodulin, ICAM-3, E-Selectin and P-Selectin) as measure by blood samples.

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego Altman Clinical & Translational Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/45/NCT04779645/ICF_000.pdf